CLINICAL TRIAL: NCT06486467
Title: Reliability of Minimally Trained Operator's Velocity-Time Integral Measurement Guided by Artificial Intelligence (MiniTrained-VTI)
Brief Title: Reliability of Minimally Trained Operator's Velocity-Time Integral Measurement Guided by Artificial Intelligence VTI
Acronym: MiniTrainedVTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Philips Healthcare (Industry); UltraSight (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: APHP230510; 2022-A02820-43 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Velocity-time Integral Measurement; Critically Ill Patients; Tissue Hypoperfusion
Keywords: Velocity-time integral; Echocardiography; Artificial Intelligence; Minimally-trained operator; Reproducibility; Fluid challenge; Fluid responsiveness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally-trained operators (Other): Group A: Minimally trained operators for LVOT VTI measurement will be intensive care residents and medical students having done less than 20 transthoracic echocardiography (TTE). All untrained operators will benefit from a standardized preliminary minimal training to teach them how to obtain apical 5-chamber view and acquire LVOT VTI using pulsed-wave Doppler according to the guidelines of the American Society of Echocardiography.
  Interventions: Other: Fluid challenge (cristalloids) OR passive leg raising
- Expert operators (Other): Group B: Experts are ICU attending physicians considered experienced and competent in TTE (either board certified or considered as experts locally). Experts will also be trained in using the same ultrasound platform equipped with the Ultrasight AI software. All operators will be trained on the same ultrasound platform: Philips Lumify® equipped with the Ultrasight AI software to optimize the quality of the 5-chamber views.
  Interventions: Other: Fluid challenge (cristalloids) OR passive leg raising

INTERVENTIONS:
Other: Fluid challenge (cristalloids) OR passive leg raising — Patients in whom fluid administration is considered necessary, based on hypoperfusion criteria will be included in the trial.
  One member of group A and one of group B will proceed independently to evaluate LVOT VTI, guided by the UltraSight AI software to obtain the best 5-chamber view. The measure of LVOT VTI will be calculated as the average of three consecutive cardiac cycles.
  The order of acquisition between group A and B will be randomized. Each operator will be blinded to the values obtained by the other.
  After baseline LVOT VTI measurement, a 250 mL fluid challenge of crystalloids or a passive leg raising test (non-pharmacological and reversible fluid challenge of roughly 250 mL), depending on the appreciation of the clinician will be performed. Measurements will be repeated immediately after the fluid challenge by the same operators, still blinded to each other, guided by the UltraSight AI software. The order of the 2nd acquisition will be the same as the 1st acquisition
  Other Names: Volume expansion

SUMMARY:
Stroke volume is a major determinant of tissue perfusion and therefore a key parameter to monitor in patients with hemodynamic instability and hypoperfusion. Left Ventricular Outflow Tract (LVOT) Velocity-Time Integral (VTI) measured using pulsed wave Doppler is widely used as an estimation of stroke volume and should be a competence required for every Intensive Care Unit (ICU) physician. Recently, research in Artificial Intelligence (AI) applied to medical imaging constituted a breakthrough in the acquisition of images. The goal of the present study is to characterize and quantify the reliability and reproducibility of LVOT VTI measurements by comparing the measures obtained by minimally-trained operators and expert physicians, guided by UltraSight AI software.

DETAILED DESCRIPTION:
The main goal of Intensive Care Unit (ICU) physicians is to ensure cellular oxygenation by maintaining adequate organ perfusion in their patients. Stroke volume is a major determinant of tissue perfusion and therefore a key parameter to monitor in patients with hemodynamic instability. Left Ventricular Outflow Tract (LVOT) Velocity-Time Integral (VTI) measured using pulsed wave Doppler is widely used as an estimation of stroke volume to assess hemodynamic modifications. This value reflects the stroke distance, which varies proportionately to stroke volume in case of hemodynamic variations resulting from therapeutic interventions (fluid administration, vasoactive drugs…) or disease processes. An increase in stroke volume (or LVOT VTI) is expected in response to fluid administration and attests for its efficacy. A lack of increase indicates that the cardiovascular system is no longer fluid-responsive, and that fluid administration is not improving tissue perfusion and creates congestion. Therefore, measuring aortic VTI should be a competence required for every ICU physician. However, international ICU guidelines on echocardiography do not consider LVOT VTI measurement as a basic skill but rather as a competence of advanced operators. More recently, the European Society of Intensive Care Medicine published expert recommendations on echocardiography, setting the evaluation of LVOT VTI as basic skill but with a weak recommendation, lacking published evidence to support this statement.

The main difficulty in measuring LVOT VTI is obtaining an adequate apical 5-chamber view.

Recently, research in artificial intelligence (AI) applied to medical imaging constituted a breakthrough in the acquisition of images. UltraSight is a company specialized in AI applied to echocardiography. Their software is based on neural network using machine learning to analyse extremely precisely the image obtained by an operator. The software indicates to the operator in real time on-screen how to optimize the image by mobilizing the probe until the desired view is correctly obtained, with the best quality.

The main objective of the present study is to characterize and to quantify the reliability and reproducibility of LVOT VTI measurements by comparing the measures obtained by minimally trained operators and experts, using an ultrasound platform equipped with real-time AI-based guidance (UltraSight). If interchangeability of minimally trained operators and expert measurements can be demonstrated, this will constitute a strong basis to upgrade the measurement of LVOT VTI as a basic competence in critical care ultrasound. The secondary objectives are to assess the concordance of therapeutic decisions made by the ICU clinician in charge of the patient (i.e.: continue or interrupt fluid administration) based on the VTI variation obtained by the minimally-trained operator, and that based on the VTI variation obtained by the expert, the agreement of the absolute value of the measure of LVOT VTI obtained by the minimally trained operators and the experts, the correlation between the measures of the VTI variation (% change following a fluid challenge of 250 mL or a passive leg-raising test) between the minimally-trained operators and those obtained by experts.

ELIGIBILITY:
Inclusion criteria:

All patients aged 18 and more

Hospitalized in ICU, in whom fluid administration is considered necessary by the clinician in charge, based on the presence of hypoperfusion criterion:

* >10% decrease in mean arterial pressure with respect to baseline value
* Skin mottling, oliguria (<0,5 ml/kg/h)
* change in the level of consciousness
* hyperlactatemia
* decrease in central venous oxygen saturation Affiliation to a French social security system (beneficiary or legal) Participant's or next of kin non-opposition or emergency procedure

Exclusion Criteria:

Patients with atrial fibrillation, due to the higher variability in LVOT VTI; Patient on Emergency Medical Assistance; Patient under guardianship, curatorship, deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative difference expressed in percentage of LVOT VTI measurement evaluated by the minimally trained operators as compared with LVOT VTI measurement by experts. | Less than 60 minutes
  To assess the equivalence of measures of LVOT VTI obtained by minimally trained operators as compared with those obtained by the experts, both guided by artificial intelligence.
  Both measures of VTI pre and post-fluid challenge will be considered.

SECONDARY OUTCOMES:
The relative difference expressed in percentage of LVOT VTI measurement, pre-fluid challenge, evaluated by the minimally trained operators as compared with those obtained by experts. | Less than 60 minutes
  To assess the equivalence of the individual measures of LVOT VTI, pre-fluid challenge, obtained by the minimally trained operators as compared with those obtained by the experts, both guided by artificial intelligence.
The relative difference expressed in percentage of LVOT VTI measurement, post-fluid challenge, evaluated by the minimally trained operators as compared with those obtained by experts. | Less than 60 minutes
  To assess the equivalence of the individual measures of LVOT VTI, post-fluid challenge, obtained by the minimally trained operators as compared with those obtained by the experts, both guided by artificial intelligence.
Difference in the VTI variation [i.e.: % change after a fluid challenge of 250 mL, or a passive leg-raising test] obtained by the minimally-trained operators and that obtained by experts. | Less than 60 minutes
  To quantify the reproducibility of LVOT VTI measurements between minimally trained operators and experts.
Correlation of the measure of the VTI variation before and after a fluid challenge of 250 mL or after a passive leg-raising test between the minimally trained operators and the experts. | Less than 60 minutes
  Correlation of the measures of the VTI variation before and after a fluid challenge of 250 mL or after a passive leg-raising test between the minimally-trained operators and the experts will be analyzed using the intraclass correlation coefficient and its associated 95% confidence interval. Pearson and Spearmann correlation coefficients will also be calculated.
Difference of the absolute value of the measure of LVOT VTI obtained by the minimally trained operators and the experts. | Less than 60 minutes
  Agreement of the absolute value of the measure of LVOT VTI obtained by the minimally trained operators and the experts using the Bland and Altman's method (bias ± limits of agreement).
Concordance in therapeutic decision by the blinded attending physician based on the measure of the VTI variation by the minimally trained operators compared to experts. | Less than 60 minutes
  Concordance in therapeutic decision by blinded attending physician (i.e.: continue or interrupt fluid administration) based on the measure of the VTI variation by the minimally trained operators compared to experts will be analyzed using the sensitivity and specificity as well as the negative and positive predictive values and its associated 95% confidence interval. The reference is the decision based on the value obtained by the expert.
Percentage of pairs (minimally-trained/expert) with difference of measurement: o < -14% o [-14%; 14%] o > 14% | Less than 60 minutes
  Percentage of pairs minimally trained/expert with difference of measurement will be described with the following thresholds:
  * < -14%
  * [-14%; 14%]
  * > 14%

CONTACTS AND LOCATIONS:
Overall Officials: Bernard MD Cholley, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - CHU de Limoges, Limoges
  - Hôpital Lariboisière - APHP, Paris
  - Hôpital européen Georges Pompidou - APHP, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR)

REFERENCES:
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Mercado P, Maizel J, Beyls C, Titeca-Beauport D, Joris M, Kontar L, Riviere A, Bonef O, Soupison T, Tribouilloy C, de Cagny B, Slama M. Transthoracic echocardiography: an accurate and precise method for estimating cardiac output in the critically ill patient. Crit Care. 2017 Jun 9;21(1):136. doi: 10.1186/s13054-017-1737-7. PMID 28595621
- [Background] Expert Round Table on Echocardiography in ICU. International consensus statement on training standards for advanced critical care echocardiography. Intensive Care Med. 2014 May;40(5):654-66. doi: 10.1007/s00134-014-3228-5. Epub 2014 Mar 11. No abstract available. PMID 24615559
- [Background] Robba C, Wong A, Poole D, Al Tayar A, Arntfield RT, Chew MS, Corradi F, Doufle G, Goffi A, Lamperti M, Mayo P, Messina A, Mongodi S, Narasimhan M, Puppo C, Sarwal A, Slama M, Taccone FS, Vignon P, Vieillard-Baron A; European Society of Intensive Care Medicine task force for critical care ultrasonography*. Basic ultrasound head-to-toe skills for intensivists in the general and neuro intensive care unit population: consensus and expert recommendations of the European Society of Intensive Care Medicine. Intensive Care Med. 2021 Dec;47(12):1347-1367. doi: 10.1007/s00134-021-06486-z. Epub 2021 Oct 5. PMID 34787687
- [Background] Mor-Avi V, Khandheria B, Klempfner R, Cotella JI, Moreno M, Ignatowski D, Guile B, Hayes HJ, Hipke K, Kaminski A, Spiegelstein D, Avisar N, Kezurer I, Mazursky A, Handel R, Peleg Y, Avraham S, Ludomirsky A, Lang RM. Real-Time Artificial Intelligence-Based Guidance of Echocardiographic Imaging by Novices: Image Quality and Suitability for Diagnostic Interpretation and Quantitative Analysis. Circ Cardiovasc Imaging. 2023 Nov;16(11):e015569. doi: 10.1161/CIRCIMAGING.123.015569. Epub 2023 Nov 13. PMID 37955139
- [Background] Jozwiak M, Mercado P, Teboul JL, Benmalek A, Gimenez J, Depret F, Richard C, Monnet X. What is the lowest change in cardiac output that transthoracic echocardiography can detect? Crit Care. 2019 Apr 11;23(1):116. doi: 10.1186/s13054-019-2413-x. PMID 30971307
- [Derived] Levy N, Meslin S, Barthelemy R, Benremily F, Bourgeois C, Bourzeix P, Chousterman B, Djadi-Prat J, Ep A, Kezar A, Laidet C, Lanoy E, Leopold V, Pereira H, Plateker O, Rivoalen AS, de Roquetaillade C, Vignon P, Bruno J, Cholley B. Reliability of minimally trained operator's left ventricular outflow tract velocity-time integral measurement guided by artificial intelligence: protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Oct 21;15(10):e105624. doi: 10.1136/bmjopen-2025-105624. PMID 41125264